CLINICAL TRIAL: NCT03411941
Title: Observational, Retrospective Study to Evaluate the Effectiveness of Intravitreal (IVT) Aflibercept Injection in Clinical Practice in naïve Patients With Neovascular Age-related Macular Degeneration (nAMD)
Brief Title: Evaluate the Effectiveness of Intravitreal (IVT) Aflibercept Injection in Clinical Practice in naïve Patients With Neovascular Age-related Macular Degeneration (nAMD)
Acronym: REALE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 18798
Record Dates: First submitted 2018-01-21; First posted 2018-01-26 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Macular Degeneration
Keywords: nAMD: neovascular Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment-naïve nAMD patients: Patient data for whom treatment with IVT aflibercept injection was initiated as first-line treatment according to the SmPC and the SERV Guideline, in treatment-naive patients with newly diagnosed of nAMD in routine clinical practice.
  Interventions: Drug: Eylea (Aflibercept, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Eylea (Aflibercept, VEGF Trap-Eye, BAY86-5321) — IVT(Intravitreal) aflibercept treatment in routine clinical practice.

SUMMARY:
There is a need to investigate the effectiveness of IVT aflibercept injection in routine clinical practice.

The aim of this study is to collect 12-month real-world clinical data from treatment-naïve nAMD patients who started first-line treatment with IVT aflibercept injection, according to the SmPC (Summary of Product Characteristics) and the SERV (Spanish Society of Retina and Vitreous) guidelines. The effectiveness of IVT aflibercept will be assessed by the changes in VA (Visual Acuity) and CRT (Central Retinal Thickness) during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged 50 years or more at aflibercept treatment initiation.
* Treatment-naïve patients with nAMD
* Patients who initated treatment with IVT aflibercept injection between 1st April 2014 to 31st May 2016
* Patients that have been decided to be treated with IVT aflibercept with a minimum treatment follow-up with IVT aflibercept injection of at least 12-months, in accordance with the approved SmPC.
* Patients who have been provided with appropriate information about the study objectives and procedures and who have given their written informed consent.

Exclusion Criteria:

* Patients who have previously been treated with anti-VEGF intravitreal injections, systemic anti-VEGF or pro-VEGF treatments, as well as other intravitreal steroids or steroid implants for the study eye.
* Patients that switched to another treatment alternative different from IVT aflibercept injection during observation period of 12 months
* Patients with another retinal disease: diabetic retinopathy, diabetic macular edema (DME), myopic choroidal neovascularization, retinal vein occlusion (RVO), central serous chorioretinopathy (CSC), angioid streaks.
* Patients with scarring, fibrosis, or atrophy involving the center of the fovea in the study eye at treatment initiation
* Patients with advanced cataract or advanced glaucoma
* Patients with presence of retinal pigment epithelial tears or rips involving the macula in the study eye prior to treatment initiation.
* Patients who do not meet the local Guideline criteria for aflibercept treatment. Contraindications listed in the SmPC must be taken into account.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include data from adult patients newly diagnosed with nAMD who initiated and maintained anti-VEGF treatment with IVT aflibercept injection in 8 Spanish centers which treat AMD patients routinely.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Mean change in VA | From baseline to month 12
  The mean change in VA from baseline (i.e. just prior to the start of treatment) to 12 months in treatment-naïve patients with nAMD in routine clinical practice in Spain.

SECONDARY OUTCOMES:
Mean change in VA | From baseline to month 6
Proportion of patients gaining 15 or more letters | At month 6 and 12
Mean change in CRT in µm (measured by OCT) | From baseline to months 6 and 12
  OCT:Optical Coherence Tomography
Presence/absence of SRF (subretinal fluid) by OCT (yes/no) | At months 6 and 12
Presence/absence of IRF (intraretinal fluid) by OCT (yes/no) | At months 6 and 12
Presence/absence of PED (pigment epithelium detachment) (measured by OCT) | At months 6 and 12
  Absence of PED: when the maximum distance between the outer border of the RPE and the inner border of the Bruch membrane is <30 μm
Presence/absence of PED Height | At months 6 and 12
  Subfoveal and 500µm nasal and temporal; PED height defined as the distance between the outer border of the retinal pigment epithelium (RPE) and the inner border of the Bruch membrane
Presence/absence of PED type | At months 6 and 12
  Serous-vascularized or fibrovascular
Correlation of the mean gain in VA with the total number of injections administered | 12 months
Mean number of IVT aflibercept injections per study eye | The first 12 months
Mean number of monitoring visits per study eye | The first 12 months
  Visits only for diagnostic/follow-up purposes, but without injections
Mean number of combined visits per study eye | The first 12 months
  Visits for monitoring and injection
Mean number of OCT assessments per study eye | The first 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many locations, Multiple Locations, Spain